CLINICAL TRIAL: NCT03376659
Title: A Phase I/II Trial of the PD-L1 Inhibitor, Durvalumab Plus CV301 in Combination With Maintenance Chemotherapy for Patients With Metastatic Colorectal or Pancreatic Adenocarcinoma
Brief Title: Durvalumab Plus CV301 With Maintenance Chemotherapy in Metastatic Colorectal or Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study closed due to lack of enrollment.
Sponsor: Georgetown University (Other)
Collaborators: Mayo Clinic (Other); Indiana University (Other); Emory University (Other); National Cancer Institute (NCI) (NIH); George Mason University (Other); Thomas Jefferson University (Other); MedImmune LLC (Industry); Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1189
Record Dates: First submitted 2017-11-20; First posted 2017-12-18 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Colorectal Cancer; Colorectal Adenocarcinoma; Pancreatic Adenocarcinoma; Metastatic Pancreatic Cancer
Keywords: PD-L1
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms | interventions — durvalumab; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I - Safety (Experimental): * MVA-BN-CV301 (prime) - Day 1 and Day 29.
  * FPV-CV301 (boost) - Day 1 of Weeks 9, 13, 17, 21, 25, 37, and q24 weeks starting week 53.
  * Durvalumab - q2 weeks
  * Capecitabine - twice a day, Monday - Friday Weekly
  * Bevacizumab - q2weeks (colorectal cancer patients only)
  Interventions: Drug: Durvalumab; Biological: CV301; Drug: Capecitabine; Drug: Bevacizumab
- Phase II - Colorectal Cancer Arm (Experimental): * MVA-BN-CV301 (prime) - Day 1 and Day 29.
  * FPV-CV301 (boost) - Day 1 of Weeks 9, 13, 17, 21, 25, 37, and q24 weeks starting week 53.
  * Durvalumab - q2 weeks
  * Capecitabine - twice a day, Monday - Friday Weekly
  * Bevacizumab - q2weeks
  Interventions: Drug: Durvalumab; Biological: CV301; Drug: Capecitabine; Drug: Bevacizumab
- Phase II - Pancreatic Cancer Arm (Experimental): * MVA-BN-CV301 (prime) - Day 1 and Day 29.
  * FPV-CV301 (boost) - Day 1 of Weeks 9, 13, 17, 21, 25, 37, and q24 weeks starting week 53.
  * Durvalumab - q2 weeks
  * Capecitabine - twice a day, Monday - Friday Weekly
  Interventions: Drug: Durvalumab; Biological: CV301; Drug: Capecitabine

INTERVENTIONS:
Drug: Durvalumab — 750mg IV q2 weeks
  Other Names: MEDI4736
Biological: CV301 — MVA-BN-CV301 (prime) - two priming doses of 1.6 x 109 infectious units/0.5 mL (Inf.U) given subcutaneously (s.c.)
  FPV-CV301 (boost) - dosed at 1 × 109 Inf.U/0.5 mL given s.c.
Drug: Capecitabine — 1000mg orally twice a day, Monday - Friday Weekly
  Other Names: Xeloda
Drug: Bevacizumab — 5mg/kg IV q2weeks
  Other Names: Avastin
  Arms: Phase I - Safety; Phase II - Colorectal Cancer Arm

SUMMARY:
This is a dual arm, open label phase I/II study to evaluate the safety and clinical activity of the combination of durvalumab with CV301 in combination with maintenance chemotherapy for patients with metastatic colorectal or pancreatic cancer whose disease is stable on, or responding to 1st line therapy for metastatic disease. Patients with metastatic colorectal or pancreatic adenocarcinoma who still have an adequate performance status and normal hepatic and renal function will be eligible.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven metastatic pancreatic or colorectal adenocarcinoma with measurable disease, defined as at least 1 unidimensionally measurable lesion on a CT scan as defined by RECIST 1.1 criteria.
2. Stable on, or responding to 1st line therapy for metastatic disease

   1. At least 8 and not more than 16 weeks after initiating 1st line therapy for metastatic disease
   2. Tumor stability/response on 1st line therapy will be determined as per RECIST 1.1
3. Prior adjuvant chemotherapy is allowed, as long as a minimum of 3 months (for pancreatic cancer) and 6 months (for colorectal cancer) has passed between the completion of adjuvant therapy and the start of first line therapy
4. Disease that is amenable to serial biopsies
5. ECOG performance status 0-1
6. Age >= 18 years
7. Blood pressure <160/100 mmHg
8. Adequate hepatic, bone marrow, and renal function:

   1. Bone Marrow: Absolute neutrophil count (ANC) ≥ 1,500/mm3; Platelets ≥ 100,000/mm3; Hemoglobin ≥ 9.0 g/dL
   2. Renal function: Serum creatinine ≤ 1.5 X upper normal limit of institution's normal range OR creatinine clearance ≥ 40 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal. Creatinine clearance should be determined by the Cockcroft-Gault formula (below) or by 24-hour urine collection for determination of creatinine clearance:

      Males:

      Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

      Females:

      Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
   3. Hepatic function: AST and ALT ≤ 2.5 X the upper normal limit of institution's normal range. Non-fasting bilirubin ≤ 1.5 X the upper normal limit of institution's normal range.
9. Partial Thromboplastin Time (PTT) must be ≤ 1.5 X upper normal limit of institution's normal range and INR (International Normalized Ratio) ≤ 1.5. Subjects on anticoagulant (such as coumadin) will be permitted to enroll as long as the INR is in the acceptable therapeutic range as determined by the investigator. Due to the drug-drug interaction between warfarin and capecitabine, alternate anticoagulation should be considered.
10. Life expectancy > 12 weeks.
11. Women of childbearing potential must have a negative serum or urine pregnancy test within 28 days prior to initiation of treatment AND confirmed prior to initiation of treatment on Day 1.
12. Alternatively, female subjects must be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy).
13. Subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consents, approved by the Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. Any prior immunotherapy or vaccine therapy
2. History of active or prior documented autoimmune disease within the past 2 years including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, auto-immune Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, with the following caveats:

   * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
   * Patients with Grave's disease, vitiligo, autoimmune alopecia, or psoriasis not requiring systemic treatment (within the past 2 years) are eligible upon consultation with the Study Chairs
   * Patients with questionable diagnosis of autoimmune disease who have never been treated with immunosuppressive regimen and have no ongoing symptoms at the time of enrollment may be eligible after discussion with medical monitor and principle investigator
3. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and TNFα antagonists) within 28 days prior to Week 1, Day 1

   * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the Study Co-chairs.
   * The use of inhaled, intranasal, ophthalmic or topical corticosteroids is allowed
   * The use of mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension is allowed.
   * Physiologic doses of systemic corticosteroids at doses which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
   * High dose steroid pre-treatment for CT contrast dye allergy is allowed, provided the dose(s) of steroids is(are) given at least 1 week prior to starting the study medications
4. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan

   o History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
5. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
6. Positive test for HIV infection
7. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening)

   o Patients with past or resolved hepatitis B infection (defined as having a negative HBsAg test and a positive IgG antibody to hepatitis B core antigen [anti-HBc] OR negative HBV viral load by PCR) are eligible.
8. Active hepatitis C

   o Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.
9. Active tuberculosis OR known history of previous clinical diagnosis of tuberculosis
10. Severe infections within 4 weeks prior to Week 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia

    o Any course of oral or IV antibiotics must have been completed at least 2 weeks prior to the first dose of study medications
11. Signs or symptoms of infection within 2 weeks prior to Week 1, Day 1
12. Received oral or IV antibiotics within 2 weeks prior to Week 1, Day 1

    o Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
13. Prior allogeneic bone marrow transplantation or prior solid organ transplantation
14. Administration of a live, attenuated vaccine within 30 days before Week 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study

    o Influenza vaccination should be given during influenza season only. Patients must not receive live, attenuated influenza vaccine (e.g., FluMistTM) within 4 weeks prior to Week 1, Day 1 or at any time during the study.
15. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
16. Any anti-cancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 2 weeks prior to initiation of study treatment, with the following exceptions:

    * Hormone-replacement therapy or oral contraceptives
    * Herbal therapy > 1 week before Week 1, Day 1 (herbal therapy intended as anti-cancer therapy must be discontinued at least 1 week before Week 1, Day 1)
17. CNS metastases including a history of leptomeningeal carcinomatosis
18. Subjects with uncontrolled seizures
19. The subject has had another active malignancy within the past five years except for cervical cancer in situ, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin. Questions regarding the inclusion of individual subjects should be directed to the Principle Investigator.
20. Cardiovascular disease including unstable angina, therapy for life-threatening ventricular arrhythmia, or myocardial infarction, stroke, or congestive heart failure within the last 6 months
21. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
22. Life-threatening visceral disease or other severe concurrent disease
23. Grade ≥2 proteinuria at screening (or known prior)
24. Women who are pregnant or breastfeeding, or male or female patients of reproductive potential who are not employing two highly effective and acceptable forms of contraception throughout their participation in the study and for 90 days after last dose of study drug.
25. Patients concurrently receiving any other investigational agents.
26. History of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab or any excipient or any egg products
27. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pishvaian, MD PhD, Study Chair — Johns Hopkins University
Locations (1):
- Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study terminated during Phase I. No subjects enrolled in Phase II.
Groups:
- Phase I - Safety- Colorectal Cancer Arm: * MVA-BN-CV301 (prime) - Day 1 and Day 29.
  * FPV-CV301 (boost) - Day 1 of Weeks 9, 13, 17, 21, 25, 37, and q24 weeks starting week 53.
  * Durvalumab - q2 weeks
  * Capecitabine - twice a day, Monday - Friday Weekly
  * Bevacizumab - q2weeks (colorectal cancer patients only)
  Durvalumab: 750mg IV q2 weeks
  CV301: MVA-BN-CV301 (prime) - two priming doses of 1.6 x 109 infectious units/0.5 mL (Inf.U) given subcutaneously (s.c.)
  FPV-CV301 (boost) - dosed at 1 × 109 Inf.U/0.5 mL given s.c.
  Capecitabine: 1000mg orally twice a day, Monday - Friday Weekly
  Bevacizumab: 5mg/kg IV q2weeks
- Phase I - Safety- Pancreatic Cancer Arm: * MVA-BN-CV301 (prime) - Day 1 and Day 29.
  * FPV-CV301 (boost) - Day 1 of Weeks 9, 13, 17, 21, 25, 37, and q24 weeks starting week 53.
  * Durvalumab - q2 weeks
  * Capecitabine - twice a day, Monday - Friday Weekly
  Durvalumab: 750mg IV q2 weeks
  CV301: MVA-BN-CV301 (prime) - two priming doses of 1.6 x 109 infectious units/0.5 mL (Inf.U) given subcutaneously (s.c.)
  FPV-CV301 (boost) - dosed at 1 × 109 Inf.U/0.5mL given s.c.
  Capecitabine: 1000mg orally twice a day,Monday - Friday Weekly
Period: Overall Study
Arm/Group | Phase I - Safety- Colorectal Cancer Arm | Phase I - Safety- Pancreatic Cancer Arm
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I - Safety- All Groups: * MVA-BN-CV301 (prime) - Day 1 and Day 29.
  * FPV-CV301 (boost) - Day 1 of Weeks 9, 13, 17, 21, 25, 37, and q24 weeks starting week 53.
  * Durvalumab - q2 weeks
  * Capecitabine - twice a day, Monday - Friday Weekly
  * Bevacizumab - q2weeks (colorectal cancer patients only)
  Durvalumab: 750mg IV q2 weeks
  CV301: MVA-BN-CV301 (prime) - two priming doses of 1.6 x 109 infectious units/0.5 mL (Inf.U) given subcutaneously (s.c.)
  FPV-CV301 (boost) - dosed at 1 × 109 Inf.U/0.5 mL given s.c.
  Capecitabine: 1000mg orally twice a day, Monday - Friday Weekly
  Bevacizumab: 5mg/kg IV q2weeks
Arm/Group | Phase I - Safety- All Groups
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose of Durvalumab
Description: The Recommended Phase II dose of durvalumab in the combination of durvalumab plus CV301 with maintenance chemotherapy as determined by the Phase I design
Time Frame: 6 months
Population: Phase 1 not completed because study terminated due to lack of enrollment. Recommended phase II dose could not be determined.
Groups:
- Phase I - Safety: * MVA-BN-CV301 (prime) - Day 1 and Day 29.
  * FPV-CV301 (boost) - Day 1 of Weeks 9, 13, 17, 21, 25, 37, and q24 weeks starting week 53.
  * Durvalumab - q2 weeks
  * Capecitabine - twice a day, Monday - Friday Weekly
  * Bevacizumab - q2weeks (colorectal cancer patients only)
  Durvalumab: 750mg IV q2 weeks
  CV301: MVA-BN-CV301 (prime) - two priming doses of 1.6 x 109 infectious units/0.5 mL (Inf.U) given subcutaneously (s.c.)
  FPV-CV301 (boost) - dosed at 1 × 109 Inf.U/0.5 mL given s.c.
  Capecitabine: 1000mg orally twice a day, Monday - Friday Weekly
  Bevacizumab: 5mg/kg IV q2weeks
Arm/Group | Phase I - Safety
Number analyzed (Participants) | 0

2. Primary Outcome: Progression Free Survival (PFS) Colorectal Cancer
Description: To determine the progression free survival (PFS) of durvalumab plus CV301 in combination with maintenance capecitabine and bevacizumab in patients with metastatic colorectal cancer, whose disease is stable on, or responding to 1st line therapy for metastatic disease
Time Frame: 24 months
Population: colorectal cancer
Measure: Median (Full Range); unit: months
Groups:
- Phase I - Safety- Colorectal Cancer: * MVA-BN-CV301 (prime) - Day 1 and Day 29.
  * FPV-CV301 (boost) - Day 1 of Weeks 9, 13, 17, 21, 25, 37, and q24 weeks starting week 53.
  * Durvalumab - q2 weeks
  * Capecitabine - twice a day, Monday - Friday Weekly
  * Bevacizumab - q2weeks (colorectal cancer patients only)
  Durvalumab: 750mg IV q2 weeks
  CV301: MVA-BN-CV301 (prime) - two priming doses of 1.6 x 109 infectious units/0.5 mL (Inf.U) given subcutaneously (s.c.)
  FPV-CV301 (boost) - dosed at 1 × 109 Inf.U/0.5 mL given s.c.
  Capecitabine: 1000mg orally twice a day, Monday - Friday Weekly
  Bevacizumab: 5mg/kg IV q2weeks
Arm/Group | Phase I - Safety- Colorectal Cancer
Number analyzed (Participants) | 4
months | 7.4 [3.2 to 12.9]

3. Primary Outcome: Progression Free Survival (PFS) Pancreatic Cancer
Description: To determine the progression free survival rate (PFS) of durvalumab plus CV301 in combination with maintenance capecitabine in patients with metastatic pancreatic cancer, whose disease is stable on, or responding to 1st line therapy for metastatic disease
Time Frame: 24 months
Population: pancreatic cancer
Measure: Median (Full Range); unit: months
Groups:
- Phase I - Safety- Pancreatic Cancer: * MVA-BN-CV301 (prime) - Day 1 and Day 29.
  * FPV-CV301 (boost) - Day 1 of Weeks 9, 13, 17, 21, 25, 37, and q24 weeks starting week 53.
  * Durvalumab - q2 weeks
  * Capecitabine - twice a day, Monday - Friday Weekly
  Durvalumab: 750mg IV q2 weeks
  CV301: MVA-BN-CV301 (prime) - two priming doses of 1.6 x 109 infectious units/0.5 mL (Inf.U) given subcutaneously (s.c.)
  FPV-CV301 (boost) - dosed at 1 × 109 Inf.U/0.5 mL given s.c.
  Capecitabine: 1000mg orally twice a day, Monday - Friday Weekly
Arm/Group | Phase I - Safety- Pancreatic Cancer
Number analyzed (Participants) | 4
months | 4.5 [2.8 to 7.3]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the proportion of patients whose best overall response recorded during treatment is either CR or PR according to the RECIST version 1.1.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Safety- All Groups
Number analyzed (Participants) | 8
Participants | 2

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from consenting to determination of tumor progression by RECIST version 1.1 or death due to any cause, whichever occurs first.
Time Frame: 24 months
Measure: Median (Full Range); unit: months
Groups:
- Phase I - Safety- Overall: * MVA-BN-CV301 (prime) - Day 1 and Day 29.
  * FPV-CV301 (boost) - Day 1 of Weeks 9, 13, 17, 21, 25, 37, and q24 weeks starting week 53.
  * Durvalumab - q2 weeks
  * Capecitabine - twice a day, Monday - Friday Weekly
  * Bevacizumab - q2weeks (colorectal cancer patients only)
  Durvalumab: 750mg IV q2 weeks
  CV301: MVA-BN-CV301 (prime) - two priming doses of 1.6 x 109 infectious units/0.5 mL (Inf.U) given subcutaneously (s.c.)
  FPV-CV301 (boost) - dosed at 1 × 109 Inf.U/0.5 mL given s.c.
  Capecitabine: 1000mg orally twice a day, Monday - Friday Weekly
  Bevacizumab: 5mg/kg IV q2weeks
Arm/Group | Phase I - Safety- Overall
Number analyzed (Participants) | 8
months | 4.7 [2.8 to 12.9]

6. Secondary Outcome: Overall Survival (OS)
Description: To determine overall survival, subjects will be followed from time of consent until death (or until study termination). Subject will be followed for survival after discontinuing study medication and after the adverse event collection period has ended.
Time Frame: 4 years
Population: number of subjects still alive at the end of the study follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Safety- All Groups
Number analyzed (Participants) | 8
Participants | 1

7. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the proportion of patients with a documented CR, PR, or SD at 4 months according to the RECIST version 1.1.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Safety- All Groups
Number analyzed (Participants) | 8
Participants | 5

8. Secondary Outcome: Tolerability and Safety of the Combination
Description: Tolerability and safety of the combination as determined by the number of patients with treatment emergent adverse events
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Safety- All Groups
Number analyzed (Participants) | 8
Participants | 8

9. Secondary Outcome: Duration of Response
Description: The duration of response will also be captured as the time from which a response was first identified, until progression of disease according to the RECIST version 1.1 (or death due to any cause).
Time Frame: 1 year
Measure: Mean (Full Range); unit: days
Arm/Group | Phase I - Safety- All Groups
Number analyzed (Participants) | 8
days | 145 [59 to 172]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were assessed from time of written informed consent is obtained through 90 days after the last dose, 2 years. All-Cause Mortality was assessed up to 4 years.
Arm/Group | Phase I - Safety
All-Cause Mortality (participants affected / at risk) | 7/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Safety (N=8)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify: Stomatitis (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) — Gum Recession
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (6)
Fever (General disorders) | 2 (2)
Injection site reaction (General disorders) | 6 (6)
Allergic Reaction (Immune system disorders) | 1 (1)
Infections and infestations - Other, specify: Influenza (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — Rt lower extremity pain
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Dysuria
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Amenorrhea (Reproductive system and breast disorders) | 1 (1)
flu like symptoms (General disorders) | 1 (1)
Pimple lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
gingival hemorrhage (Gastrointestinal disorders) | 1 (1)
left upper arm mass (General disorders) | 1 (1)
oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Gingival Pain (Gastrointestinal disorders) | 1 (1)
Lipase Increased (Investigations) | 1 (3)
Paresthesia (Nervous system disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03376659/Prot_SAP_000.pdf